CLINICAL TRIAL: NCT04114604
Title: Respiratory Capacity and Swallowing Function in Spinal Disorders: A Pilot Study
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-6310; 5R01DC011020 (NIH); CAPCR 16-6310 (Other: UHN Research Ethics Board)
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries; Deglutition Disorders
MeSH Terms: conditions — Spinal Cord Injuries; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spinal Cord Injury: Adults who have sustained a spinal cord injury at the cervical or upper thoracic level (T6 or higher).

SUMMARY:
This study is part of a larger grant, for which the overall goal is to collect measurements of liquid flow through the oropharynx (i.e., mouth and throat) during swallowing.The focus of this study is to evaluate the flow of liquids of varying consistency in the spinal disorder population.

DETAILED DESCRIPTION:
Thickened liquids are commonly used as an intervention for dysphagia (swallowing impairment). However, the field lacks a clear understanding of how liquids of different consistencies behave during swallowing. In order to improve understanding of the effectiveness of altered liquid consistency for improving dysphagia, the investigators are studying liquid flow through the oropharynx. This study explores this question in individuals with spinal cord injury. Participants will swallow 20% w/v barium thickened to different consistencies (thin, slightly thick, mildly thick, moderately thick and extremely thick). Swallowing will be observed under videofluoroscopy. Simultaneous measures of airflow via nasal cannula will be used to study respiratory-swallow coordination in this study sample.

ELIGIBILITY:
Inclusion Criteria:

Spinal cord injury at the cervical or thoracic level (T6 or higher)

Exclusion Criteria:

* Prior history of swallowing, motor speech, gastro-esophageal difficulties, chronic sinusitis or taste disturbance.
* Neurological difficulties unrelated to spinal disorder (e.g. Stroke, Parkinson disease, etc).
* Cognitive communication difficulties that may hinder ability to participate.
* Current use of mechanical ventilation
* External instrumentation around the head/neck that would obstruct the field of view during the videofluoroscopy exam (e.g. cervical collar).
* Type 1 Diabetes (due to the requirement to swallow stimuli containing starch based thickeners, which carry a significant carbohydrate load).
* Known allergies to latex, food coloring or dental glue (due to the probability that these items will come into contact with the oral mucosa during data collection).
* Children and pregnant women (due to the use of radiation during the videofluoroscopic examination).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit participants from the inpatient SCI program at the Toronto Rehabilitation Institute Lyndhurst Center.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Steele, Principal Investigator — KITE - Toronto Rehabilitation Institute, University Health Network
Locations (1):
- Toronto Rehabilitation Institute - Lyndhurst Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
not planned at this time

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spinal Cord Injury
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Injury
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 49 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Displaying Unsafe Swallowing
Description: The Penetration-Aspiration Scale is an 8-point categorical scale that is used to characterize swallowing safety for each bolus based on the depth to which any material enters the airway and whether or not the material is ejected. Levels 1 and 2 on the scale are considered safe, while levels > 2 are considered unsafe. Actual scale scores (1-8) will be recorded and then converted to binary categorical scores (< 3 vs >/= 3). We report the frequency (count) of participants showing unsafe swallowing (i.e., scores > 2) by bolus consistency.
Time Frame: Baseline (single timepoint only)
Population: Adults who have sustained a spinal cord injury at the cervical or upper thoracic level (T6 or higher).
Measure: Count of Participants; unit: Participants
Groups:
- Thin Liquid Barium: Participants were asked to take a series of 3 comfortable sips of thin liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque powder and water.
- Slightly Thick Liquid Barium: Participants were asked to take a series of 3 comfortable sips of slightly thick liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque powder, water and Nestle Resource ThickenUp Clear thickener.
- Mildly Thick Liquid Barium: Participants were asked to take a series of 3 comfortable sips of mildly thick liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque powder, water and Nestle Resource ThickenUp Clear thickener.
- Moderately Thick Liquid Barium: Participants were asked to take a series of 3 comfortable sips of moderately thick liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque powder, water and Nestle Resource ThickenUp Clear thickener.
- Extremely Thick Liquid Barium: Participants were asked to take a series of 3 comfortable sips of extremely thick liquid barium prepared in 20% w/v concentration using Bracco E-Z-Paque powder, water and Nestle Resource ThickenUp Clear thickener.
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Displaying Post-swallow Inhalation
Description: Healthy swallowing typically occurs partway through an outward breath, such that the direction of breathing both before and after the swallow is exhalation. Whenever a swallow is followed immediately by inhalation, this is considered abnormal and a risk for food or liquid material to be sucked into the airway. We measured the direction of breathing before and after swallows via nasal cannula using the airflow module of the KayPentax Digital Swallow Workstation Swallowing Signals Lab. We report the frequency (percentage) of participants displaying at least one swallow showing post-swallow inhalation by consistency.
Time Frame: Baseline (single timepoint only)
Population: A sample of 10 adults was enrolled. Due to signal quality issues, data were missing for one participant across all consistencies and for an additional participant on moderately thick liquid barium.
Measure: Count of Participants; unit: Participants
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
Participants | 2 | 5 | 3 | 1 | 2

3. Primary Outcome: Duration of the Respiratory Pause Seen in Swallowing
Description: Healthy swallowing typically occurs partway through an outward (exhalatory) breath, and involves a pause in breathing. The duration of this respiratory pause was measured in milliseconds for each swallow based on the continuous airflow waveform collected via nasal cannula using the airflow module of the KayPentax Digital Swallow Workstation Swallowing Signals Lab. We report means and standard deviations for respiratory pause duration by consistency. Shorter respiratory pause durations reflect inadequate airway protection.
Time Frame: Baseline (single timepoint only)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Thin Liquid Barium | Slightly Thick Liquid Barium | Mildly Thick Liquid Barium | Moderately Thick Liquid Barium | Extremely Thick Liquid Barium
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 9
milliseconds | 901 (485) | 996 (573) | 867 (455) | 721 (275) | 815 (541)

ADVERSE EVENTS:
Time Frame: 1 week following data collection
Arm/Group | Spinal Cord Injury
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04114604/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT04114604/ICF_001.pdf